CLINICAL TRIAL: NCT07332585
Title: Efficacy of Piezosurgery Versus Conventional Osteotomy in Prelacrimal Approach Targeting Different Maxillary Sinus Pathologies: a Randomized Controlled Trial
Brief Title: Efficacy of Piezosurgery Versus Conventional Osteotomy in Prelacrimal Approach Targeting Different Maxillary Sinus Pathologies
Acronym: prelacrimal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.24.11.2964
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Maxillary Sinus Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- piezosurgery group (Active Comparator)
  Interventions: Procedure: piezo-assisted prelacrimal apporach
- conventional osteotomy group (Active Comparator)
  Interventions: Procedure: conventional osteotomy prelacrimal approach

INTERVENTIONS:
Procedure: piezo-assisted prelacrimal apporach — The removal of the bone in the prelacrimal approach was done using piezo ultrasonic device
  Arms: piezosurgery group
Procedure: conventional osteotomy prelacrimal approach — The removal of the bone in the prelacrimal approach was done using conventional osteotome and hammer
  Arms: conventional osteotomy group

SUMMARY:
The prelacrimal recess approach is a minimally invasive approach to maxillary sinus lesions. The current study aimed to evaluate the efficacy of piezosurgery versus conventional osteotomy while performing a prelacrimal apporach.

ELIGIBILITY:
Inclusion Criteria:

1. Any maxillary sinus pathology (recurrent Antrochoanal polyp, inverted papilloma, fungal ball, allergic fungal sinusitis, CRSwNP, CRSeNP, orbital floor fracture, etc).
2. Favorable prelacrimal recess (Type II or III Simmen classification)
3. Age> 18 years.
4. No gender limitation.

Exclusion Criteria:

1. patients with malignant sino-nasal tumors.
2. patients unfit for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative bleeding | During the surgical procedure
  The amount of blood collected in the suction device
Operative time | During the surgical procedure
  the time of surgical procedure

SECONDARY OUTCOMES:
Postoperative hyposthesia | six months after surgery
  hyposthesia in the cheek and upper teeth after surgery, measured by the Barrow Institution grading of hyposthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt